CLINICAL TRIAL: NCT00708461
Title: Environmental Intervention for Weight Gain Prevention
Acronym: HealthWorks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0408S62609; 5R01DK067362 (NIH)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity
Keywords: obesity; obesity prevention; worksite; environment; intervention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Worksite Environmental Intervention (Experimental): Changes to healthy food availability, physical activity opportunities and promotion, body weight scale access, and media enhancements to target weight gain prevention
  Interventions: Behavioral: weight gain prevention
- No-contact control (No Intervention): No-treatment control condition. Worksites were offered program materials upon completion of programs at intervention sites.

INTERVENTIONS:
Behavioral: weight gain prevention — 1. Changes in the food environment that increase the availability of healthy foods and beverages, reduce food and beverage portion sizes, reduce prices on healthy food items, and increase prices on less healthy food items.
  2. Changes in the activity environment that increase cues and incentives for walking at work and at home, using stairs, and to increase exposure of employees to information about active recreational opportunities at work and at home.
  3. Changes to the environment to increase cues and incentives for regular weight monitoring by providing scales at convenient locations.
  4. Changes in the informational environment that increase frequency of exposure of the employee population to accurate information about healthy food and activity choices.
  Other Names: worksite intervention; obesity prevention
  Arms: Worksite Environmental Intervention

SUMMARY:
The primary aim of this research is to evaluate the efficacy of a multicomponent worksite-based, environmental intervention in reducing weight increase and obesity over time in working adults.

DETAILED DESCRIPTION:
This study is a randomized trial designed to evaluate the effectiveness of a multi-component worksite intervention with strong environmental components to prevent weight gain. Six worksites will be randomized to either an intervention or a no-treatment control group. The intervention will be comprised of 1) changing the availability, portion sizes, and prices of foods and beverages sold to employees in their worksites in ways that encourage healthier food choices; 2) increasing the availability of physical activity opportunities at the worksite by implementing walking programs and increasing stairwell access and attractiveness; 3) placing scales in the work environment to encourage body weight monitoring and to enable workers to set goals for their weight; and 4) to provide educational materials to all employees to make them aware of the environmental intervention and of behavioral practices likely to be effective in preventing weight gain. The intervention will be implemented for a 2-year period in each intervention site. Effectiveness will be evaluated by assessing body weight, eating behavior and physical activity in a cohort of employees in both control and intervention sites at baseline and again 2 years later. Weight trends in these populations will also be compared to data from national and state-level annual surveys of weight in representative population samples. Data will be collected on the effects of specific intervention components via aggregate measures of food choice and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* generally in good health
* part- or full-time employee in one of the participating worksites

Exclusion Criteria:

* work on site <50% of the time
* work second or third shift

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1747 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Jeffery, PhD, Principal Investigator — University of Minnesota, Division of Epidemiology and Community Health
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] VanWormer JJ, Linde JA, Harnack LJ, Stovitz SD, Jeffery RW. Weight change and workplace absenteeism in the HealthWorks study. Obes Facts. 2012;5(5):745-52. doi: 10.1159/000345119. Epub 2012 Oct 24. PMID 23108493
- [Result] Linde JA, Nygaard KE, MacLehose RF, Mitchell NR, Harnack LJ, Cousins JM, Graham DJ, Jeffery RW. HealthWorks: results of a multi-component group-randomized worksite environmental intervention trial for weight gain prevention. Int J Behav Nutr Phys Act. 2012 Feb 16;9:14. doi: 10.1186/1479-5868-9-14. PMID 22340088
- [Result] VanWormer JJ, Linde JA, Harnack LJ, Stovitz SD, Jeffery RW. Is baseline physical activity a determinant of participation in worksite walking clubs? Data from the HealthWorks Trial. J Phys Act Health. 2012 Aug;9(6):849-56. doi: 10.1123/jpah.9.6.849. Epub 2011 Jul 29. PMID 21952267
- [Result] VanWormer JJ, Linde JA, Harnack LJ, Stovitz SD, Jeffery RW. Self-weighing frequency is associated with weight gain prevention over 2 years among working adults. Int J Behav Med. 2012 Sep;19(3):351-8. doi: 10.1007/s12529-011-9178-1. PMID 21732212
- [Derived] Graham DJ, Linde JA, Cousins JM, Jeffery RW. Environmental modifications and 2-year measured and self-reported stair-use: a worksite randomized trial. J Prim Prev. 2013 Dec;34(6):413-22. doi: 10.1007/s10935-013-0323-2. PMID 23979097
- See also: HealthWorks is a study housed in the University of Minnesota Obesity Prevention Center. — http://www.ahc.umn.edu/opc/research/OPC_Currently_Funded/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at worksites between January 2006 and April 2007. Human resources departments provided worksite contact information for all eligible employees; these email addresses and phone numbers were used for recruitment contact purposes.
Pre-assignment Details: A company-wide email was sent to eligible employees at all sites, describing the study and the partnership with the University. Employees were notified that a study staff member would contact them about the project within the next two weeks and were given the option to call study staff in advance to opt out or to enroll in the study.
Period: Overall Study
Arm/Group | Worksite Environmental Intervention | No-contact Control
Started | 752 | 995
Completed | 611 | 795
Not Completed | 141 | 200
Not completed — Lost to Follow-up | 18 | 11
Not completed — Withdrawal by Subject | 8 | 9
Not completed — left workforce | 115 | 180

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Worksite Environmental Intervention | No-contact Control | Total
Number analyzed (Participants) | 752 | 995 | 1747
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 32 | 49
  Between 18 and 65 years | 729 | 954 | 1683
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (10.8) | 43.1 (10.6) | 42.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 478 | 608 | 1086
  Male | 274 | 387 | 661
Region of Enrollment [Number; unit: participants]
  United States | 752 | 995 | 1747

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (BMI)
Description: Assessed in kilograms per meter squared.
Time Frame: Baseline to 24 months
Population: Participants with complete data at baseline and two years, and those who were not pregnant at either time, were retained for analysis.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared
Arm/Group | Worksite Environmental Intervention | No-contact Control
Number analyzed (Participants) | 580 | 742
kilograms per meter squared | 0.315 (0.08959) | 0.190 (0.07987)
Statistical Analysis 1: Comparison: Worksite Environmental Intervention vs No-contact Control; The null hypothesis was no effect of the environmental intervention. The following power assumptions were made: * Intraclass correlation (ICC) of 0.016, estimated from an earlier study * Variance of 118 kg, estimated from an earlier study * Cohort N=400 * 15% attrition (by turnover) Using the external control and a worksite correlation of 0.2 gives a detectable difference of about 1.5 kg or 3 lb, or an effect size of 0.14. The effect size using internal control is 0.20; Test type: Superiority or Other; p = 0.36, ANCOVA — Adjusted for age, educational attainment, race/ethnicity, and smoking status as individual, fixed-effect covariates. 95% confidence intervals and p-values derived from t-statistics with 4 degrees of freedom, reflecting the group-randomized design; Adjusted for age, educational attainment, race/ethnicity, and smoking status as individual, fixed-effect covariates; Mean Difference (Net) = 0.125, 95% CI 2-sided [-0.21 to 0.46], Standard Error of Mean 0.1202

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for the duration of the study (2 years at each site).
Arm/Group | Worksite Environmental Intervention | No-contact Control
Serious Adverse Events (participants affected / at risk) | 0/752 | 0/995
Other Adverse Events (participants affected / at risk) | 0/752 | 0/995

LIMITATIONS AND CAVEATS:
The recruitment goal of 6 sites represents only 3% of those initially contacted for participation, or 16% of eligible and interested sites. The design limits power due to the small sample size at the group level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No